CLINICAL TRIAL: NCT04397055
Title: Comparison of Blood Lipids From Diets Enriched With Cottonseed Oil Versus Olive Oil in Adults With High Cholesterol
Brief Title: Oil Consumption and Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: National Cottonseed Products Association (Unknown); Cotton Incorporated (Unknown); University of Georgia Obesity Initiative (Unknown)
Responsible Party: Principal Investigator, Jamie Cooper, PhD, Associate Professor, Dept. of Foods and Nutrition, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00005869
Record Dates: First submitted 2020-04-30; First posted 2020-05-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Cottonseed Oil; Olive Oil

STUDY DESIGN:
Intervention Model Description: 8 week parallel feeding trials of diets rich in Cottonseed oil or Olive Oil
Who Masked: Participant
Masking Description: Participants are blinded to which oil they are receiving
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cottonseed Oil (Experimental): Participants are given foods enriched with cottonseed oil and instructed on how to substitute study foods into their diet to maintain caloric balance
  Interventions: Dietary Supplement: Cottonseed Oil
- Olive Oil (Active Comparator): Participants are given foods enriched with olive oil and instructed on how to substitute study foods into their diet to maintain caloric balance
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Dietary Supplement: Cottonseed Oil — Participants are provided about 60% of their required energy for 8 weeks as foods from a 5 day cycle menu that are enriched with Cottonseed Oil
  Arms: Cottonseed Oil
Dietary Supplement: Olive Oil — Participants are provided about 60% of their required energy for 8 weeks as foods from a 5 day cycle menu that are enriched with Olive Oil
  Arms: Olive Oil

SUMMARY:
More than 31 million U.S. adults have high total cholesterol and over 73 million U.S. adults have high LDL cholesterol. Cottonseed oil (CSO) is found readily in our food supply, and recent research has shown improvements in blood lipids following CSO consumption in healthy adults with normal cholesterol profiles. To date, however, there are no published studies on the effects of CSO-enriched diets on blood lipids and markers of health in an older population with hypercholesterolemia. Therefore, the purpose of this study is to test the health effects of a diet rich in CSO against a diet rich in olive oil to determine if the CSO-enriched diet will show greater improvements in blood lipids and other health markers in adults with high cholesterol levels. If CSO in the diet is found to improve these markers, these study findings could lead to improvements in health.

DETAILED DESCRIPTION:
This was a single-blind, randomized controlled trial. Investigators recruited subjects with hypercholesterolemia (high blood cholesterol levels). Subjects were randomized into one of two groups: (1) Cottonseed oil (CSO), (2) Olive oil (OO). The interventions consist of identical foods that are only different in the respective oil they are prepared with.

There was a screening visit and 3 testing visits: Baseline (visit 2), mid-visit at week 4 (visit 6), and post-visit at week 8 (visit 10). Anthropometrics, questionnaires, and a fasting blood sample were collected at each visit. At visits 2 and 10 participants participated in a saturated fatty acid meal challenge in which additional blood and metabolism measurements were collected. Visits 3-9 represent weekly meal pickups, with the exception of visit 6 which is also a testing visit.

Hypothesis: Investigators hypothesized that enrichment of the diet with CSO would result in significantly greater improvements in blood lipids, metabolism, and appetite compared to the OO group.

ELIGIBILITY:
Inclusion Criteria:

* 30-75 year old
* body mass index (BMI) between 18.5-39.9 kg/m2
* higher cholesterol levels indicated by "At Risk/Borderline High" in two or more of the variables (total cholesterol: 180-239 mg/dL, LDL cholesterol 110-159 mg/dL, triglycerides 130-199 mg/dL) or "High" in either total cholesterol (240 mg/dL and higher) or LDL (160 mg/dL or higher), and having triglyceride levels less than 350mg/dL.

Exclusion Criteria:

* participants with familial hypercholesterolemia
* LDL levels greater than the 95th percentile based on age and sex
* HDL levels lower than the 20th percentile based on age and sex
* women on hormone replacement therapy for less than 2 years
* individuals who regularly exercise more than 3 h/w
* weight gain or loss more than 5% of their body weight in the past 3 months
* plans to begin a weight loss/exercise regiment during the trial
* history of medical or surgical events that could affect digestion or swallowing
* gastrointestinal surgeries
* conditions or disorders
* any chronic or metabolic diseases
* atherosclerosis
* previous MI or stroke
* cancer
* fasting blood glucose levels greater than 126 mg/dL
* blood pressure greater than 180/120 mmHg
* medication use affecting digestion and absorption
* medication use affecting metabolism (e.g. thyroid meds)
* lipid-lowering medications
* medications for diabetes
* steroid/hormone therapies
* a medically prescribed or special diet
* food allergies (specific for the foods made in the study)
* taking fish oil and calciumfloroboron supplements
* excessive alcohol use (greater than 3 drinks/d for men; greater than 2 drinks/d for women)
* tobacco or nicotine use

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Change in baseline fasting blood lipids at weeks 4 and 8 | Baseline, 4 weeks, 8 weeks
  Total Cholesterol (mg/dL), high-density lipoprotein (HDL) cholesterol (mg/dL), triglycerides (mg/dL), low-density lipoprotein (LDL) cholesterol (mg/dL), apolipoprotein B (mg/dL)
Change in baseline lipoprotein (a), lipoprotien particle number and size at weeks 4 and 8 | Baseline, 4 weeks, 8 weeks
  Low density lipoprotien (LDL) particle number (nmol/L), LDL small (nmol/L), HDL large (nmol/L), LDL medium (nmol/L), lipoprotein (a) (nmol/L).
Change in baseline low density lipoprotien (LDL) peak size at weeks 4 and 8 | Baseline, 4 weeks, 8 weeks
  LDL peak size (angstrom)

SECONDARY OUTCOMES:
Change in Baseline Blood Concentration of Hunger and Satiety Hormones over 8 weeks | measured at weeks 1 and 8 at fasting and for 5 hours postprandially
  Blood samples will be collected to measure Peptide tyrosine tyrosine (YY) (pg/mL), Cholecystokinin (CCK) (pg/mL), Ghrelin (pg/mL), Glucagon-like peptide 1 (GLP1) (pg/mL)
Change in Height over 8 weeks | measured at weeks 1, 4, and 8 at fasting
  Height measured in centimetres
Change in weight over 8 weeks | measured at weeks 1, 4, and 8 at fasting
  weight measured in pounds and kilograms
change in blood pressure over 8 weeks | measured at weeks 1, 4, and 8 at fasting
  both systolic and diastolic blood pressure measured in millimetres of mercury (mmHg)
change in waist circumference over 8 weeks | measured at weeks 1, 4, and 8 at fasting
  waist circumference measured in centimetres
change in hip circumference over 8 weeks | measured at weeks 1, 4, and 8 at fasting
  hip circumference measured in centimetres
change in total body fat percentage over 8 weeks | measured at weeks 1, 4, and 8 at fasting
  total body fat percentage measured as percent of total body mass
change in Blood glucose concentration responses (glycemia) over 8 weeks | measured at week 1 and 8 at fasting and for 5 hours postprandially
  blood samples are collected to measure blood glucose concentration (mg/dL) in response to saturated fatty acid meal
change in Blood insulin concentration responses (glycemia) over 8 weeks | measured at week 1 and 8 at fasting and for 5 hours postprandially
  blood samples are collected to measure blood insulin concentration (uU/mL) in response to saturated fatty acid meal
change in blood triglyceride meal responses over 8 weeks | measured at week 1 and 8 at fasting and for 5 hours postprandially
  Triglyceride (mg/dL) response to saturated fatty acid meal
change in non-esterified free fatty acid (NEFA) meal responses over 8 weeks | measured at week 1 and 8 at fasting and for 5 hours postprandially
  NEFA (mEq/dL) response to saturated fatty acid meal
change in Fat oxidation over 8 weeks | measured at week 1 and 8 at fasting and for 3.5 hours postprandially
  measured (g/hr) via indirect calorimetry
change in Carbohydrate oxidation over 8 weeks | measured at week 1 and 8 at fasting and for 3.5 hours postprandially
  measured (g/hr) via indirect calorimetry
change in Resting metabolic rate (RMR) over 8 weeks | measured at week 1 and 8 at fasting and for 3.5 hours postprandially
  RMR (kcals/d) measured via indirect calorimetry
change in Respiratory exchange ratio (RER) over 8 weeks | measured at week 1 and 8 at fasting and for 3.5 hours postprandially
  measured (VCO2/Vo2) via indirect calorimetry
change in subjective appetite over 8 weeks | measured at week 1 and 8 at fasting and for 5 hours postprandially in 30 minuet intervals; also measured once per hour after the subject leaves the lab until they go to bed
  hunger, fullness, prospective consumption, and desire to eat measured via a Visual Analog Scale (VAS). VAS uses an unmarked 10 centimetre line and asks the subject to answer the connected question by placing a tick mark on the line as though it is a spectrum from 0 to 100 percent with the right being in the most agreement (i.e. extremely hungry in response to how hungry are you) and the left being the most disagreement (i.e. extremely not hungry in response to how hungry are you). Answers will be measured in centimetres in response to questions about hunger, fullness, prospective consumption, and desire to eat.

OTHER OUTCOMES:
Change in Perceived Stress over 8 weeks | measured at week 1, 4, and 8 at fasting
  perceived Stress Scale is a questionnaire asking 10 questions about the subject's feelings of stress in the past month. There are 5 possible answers, never, almost never, sometimes, fairly often, very often with corresponding scores of 0 - 4 respectively. Scores for all questions will be added up as in indication of stress level. Higher perceived stress scale scores correspond to higher stress levels.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The plan is to share group averages through publication

REFERENCES:
- [Derived] Prater MC, Scheurell AR, Paton CM, Cooper JA. Eight weeks of daily cottonseed oil intake attenuates postprandial angiopoietin-like proteins 3 and 4 responses compared to olive oil in adults with hypercholesterolemia: A secondary analysis of a randomized clinical trial. Nutr Res. 2024 Mar;123:88-100. doi: 10.1016/j.nutres.2024.01.006. Epub 2024 Jan 12. PMID 38295507
- [Derived] Prater MC, Scheurell AR, Paton CM, Cooper JA. Hunger and satiety responses to diets enriched with cottonseed oil vs. olive oil. Physiol Behav. 2023 Feb 1;259:114041. doi: 10.1016/j.physbeh.2022.114041. Epub 2022 Nov 24. PMID 36427543
- [Derived] Prater MC, Scheurell AR, Paton CM, Cooper JA. Metabolic responses to 8 weeks of consuming cottonseed oil versus olive oil in adults with dyslipidaemia: a randomised trial. J Hum Nutr Diet. 2023 Jun;36(3):1079-1089. doi: 10.1111/jhn.13085. Epub 2022 Sep 16. PMID 36056703
- [Derived] Prater MC, Scheurell AR, Paton CM, Cooper JA. Blood Lipid Responses to Diets Enriched with Cottonseed Oil Compared With Olive Oil in Adults with High Cholesterol in a Randomized Trial. J Nutr. 2022 Sep 6;152(9):2060-2071. doi: 10.1093/jn/nxac099. PMID 35511204